CLINICAL TRIAL: NCT02512965
Title: A Randomized Phase II/III Study Comparing Stereotactic Body Radiotherapy(SBRT) Versus Conventional Palliative Radiotherapy (CRT) for Patients With Spinal Metastases
Brief Title: Study Comparing Stereotactic Body Radiotherapy vs Conventional Palliative Radiotherapy (CRT) for Spinal Metastases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Trans Tasman Radiation Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SC24
Record Dates: First submitted 2015-07-27; First posted 2015-07-31 (Estimated); Results first posted 2021-08-16 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2021-08

CONDITIONS: Spinal Metastases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Conventional Radiotherapy (Active Comparator): Standard Conventional Radiotherapy (CRT) 20 Gy in 5 fractions
  Interventions: Radiation: 20 Gy in 5 fractions
- Stereotactic Body Radiotherapy (Experimental): Stereotactic Body Radiotherapy (SBRT) 24 Gy in 2 fractions
  Interventions: Radiation: Conventional SBRT: 24 Gy in 2 fractions

INTERVENTIONS:
Radiation: 20 Gy in 5 fractions
  Arms: Standard Conventional Radiotherapy
Radiation: Conventional SBRT: 24 Gy in 2 fractions
  Arms: Stereotactic Body Radiotherapy

SUMMARY:
The purpose of this study is to find out if SBRT is better than CRT at controlling pain in the spine 3 months after receiving treatment.

DETAILED DESCRIPTION:
This research is being done because while there is some evidence suggesting that SBRT may improve treatment for patients with spine metastases, more research is needed to determine if it is better than CRT. The first part of the randomized trial (phase II) looked at whether it was possible (feasible) to provide these treatments in cancer centres across Canada, by aiming to recruit 54 participants within 18 months. This part of the study was successfully completed in early 2017. The second component of this study, called a randomized phase III trial, is now underway. It involves recruiting another 124 participants to receive either CRT or SBRT, using the same study procedure as in the feasibility study. We will continue to obtain information about whether SBRT is better than CRT at controlling pain.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of cancer (excluding seminoma, small cell lung cancer and hematologic primaries).
* Spinal metastasis documented with MRI and suitable for treatment with radiotherapy with the following characteristics:

  * Painful, as defined by a pain score ≥ 2 for worst pain in the planned target treatment volume;
  * ≤ 3 consecutive spinal segments involved by tumour to be included in the planned target volume. The patient may have other spinal metaastases to be treated as per the radiation oncologist's discretion, but the eligible spinal metastatic site has to be one where there is pain and no more than 3 consecutive segments to be included as clinical target volume and appropriate for either 20 Gy in 5 fractions or 24 Gy in 2 fractions per the randomization.
* There is no plan to change the pain medication on the first day of protocol treatment with radiotherapy.
* ECOG Performance Status 0-2.
* Seen by a radiation oncologist and judged to be appropriate for participation in this study including ability to tolerate protocol radiotherapy (SBRT or CRT).
* Age of 18 years or older.
* Patient is able and willing to complete the Patient Diary (pain and analgesic use).
* Patient is able (i.e. sufficiently fluent) and willing to complete the quality of life questionnaire in either English or French. The baseline assessment must be completed within required timelines, prior to randomization. Inability (illiteracy in English or French, loss of sight, or other equivalent reason) to complete the questionnaires will not make the patient ineligible for the study. However, ability but unwillingness to complete the questionnaires will make the patient ineligible.
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrollment in the trial to document their willingness to participate.
* Patients must be accessible for treatment and follow-up. Investigators must assure themselves the patients randomized on this trial will be available for complete documentation of the treatment, adverse events, and follow-up.
* In accordance with CCTG policy, protocol treatment is to begin within 3 weeks of patient randomization. From the time of successful treatment planning, no more than 12 days can elapse before the first fraction of radiotherapy is delivered.
* Women/men of childbearing potential must have agreed to use a highly effective contraceptive method. A woman is considered to be of "childbearing potential" if she has had menses at any time in the preceding 12 consecutive months. In addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation, or vasectomy/vasectomized partner. However, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures.
* Women of childbearing potential will have a pregnancy test to determine eligibility as part of the Pre-Study Evaluation; this may include an ultrasound to rule-out pregnancy if a false-positive is suspected. For example, when beta-human chorionic gonadotropin is high and partner is vasectomized, it may be associated with tumour production of hCG, as seen with some cancers. Patient will be considered eligible if an ultrasound is negative for pregnancy.

Exclusion Criteria:

* Patients who have a pacemaker, such that MRI cannot be performed or treatment cannot be delivered safely.
* Patients with prior treatment with any radionuclide within 30 days prior to randomization.
* Patients with prior radiation to the spinal segment intended to be treated with protocol radiotherapy such that the protocol therapy cannot be delivered as intended.
* Patients with prior surgery to the spinal segment intended to be treated with protocol radiotherapy.
* Patients who have received chemotherapy within 1 week prior to administration of protocol radiotherapy or who are expected/planned to receive chemotherapy within one week of completing protocol radiotherapy. Centre guidelines regarding administration of targeted non-cytotoxic therapy must be followed with the proviso that no systemic anticancer therapy should be administered within 24 hours prior to and post-radiotherapy. Endocrine therapy may be administered during radiotherapy as per the discretion of the treating physician.
* Patients with spine instability as judged by a Spinal Instability Neoplastic Score (SINS) of more than 12.
* Patients with symptomatic spinal cord compression or cauda equina syndrome resulting from bony compression or epidural compression of the spinal cord and cauda equina, respectively. Symptomatic refers to neurolic deficit in the form of motor, bowel or bladder dysfunction.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2021-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arjun Sahgal, Study Chair — Odette Cancer Centre, Sunnybrook Health Sciences Centre, Toronto ON
Locations (22):
- Australia (8):
  - Auckland City Hospital, Grafton, Aucklund
  - Liverpool Cancer Therapy Centre, Liverpool Hospital, Liverpool, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Peter McCallum Cancer Institute, Melbourne, Victoria
  - Peter Mac - Sunshine Hospital, St Albans, Victoria
  - Canberra Hospital, Garran
  - Royal Brisbane and Womens Hospital, Herston
- Canada (14):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Centre for the North, Prince George, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - BCCA - Vancouver Island Cancer Centre, Victoria, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - CHUM-Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - CHUQ-Pavillon Hotel-Dieu de Quebec, Québec, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sahgal A, Myrehaug SD, Siva S, Masucci GL, Maralani PJ, Brundage M, Butler J, Chow E, Fehlings MG, Foote M, Gabos Z, Greenspoon J, Kerba M, Lee Y, Liu M, Liu SK, Thibault I, Wong RK, Hum M, Ding K, Parulekar WR; trial investigators. Stereotactic body radiotherapy versus conventional external beam radiotherapy in patients with painful spinal metastases: an open-label, multicentre, randomised, controlled, phase 2/3 trial. Lancet Oncol. 2021 Jul;22(7):1023-1033. doi: 10.1016/S1470-2045(21)00196-0. Epub 2021 Jun 11. PMID 34126044
- [Derived] Tseng CL, Soliman H, Myrehaug S, Lee YK, Ruschin M, Atenafu EG, Campbell M, Maralani P, Yang V, Yee A, Sahgal A. Imaging-Based Outcomes for 24 Gy in 2 Daily Fractions for Patients with de Novo Spinal Metastases Treated With Spine Stereotactic Body Radiation Therapy (SBRT). Int J Radiat Oncol Biol Phys. 2018 Nov 1;102(3):499-507. doi: 10.1016/j.ijrobp.2018.06.047. Epub 2018 Jul 10. PMID 30003994

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Conventional Radiotherapy: Standard Conventional Radiotherapy (CRT) 20 Gy in 5 fractions
  20 Gy in 5 fractions
- Stereotactic Body Radiotherapy: Stereotactic Body Radiotherapy (SBRT) 24 Gy in 2 fractions
  Conventional SBRT: 24 Gy in 2 fractions
Period: Overall Study
Arm/Group | Standard Conventional Radiotherapy | Stereotactic Body Radiotherapy
Started | 115 | 114
Completed | 115 | 110 (4 patients did not receive any dose of the assigned treatment.)
Not Completed | 0 | 4
Not completed — Withdrawal by Subject | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Conventional Radiotherapy | Stereotactic Body Radiotherapy | Total
Number analyzed (Participants) | 115 | 114 | 229
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.05 (12.7) | 63.67 (12.1) | 63.86 (12.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 55 | 109
  Male | 61 | 59 | 120
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 103 | 102 | 205
  Australia | 12 | 12 | 24
ECOG Performance Status [Count of Participants; unit: Participants] — 0: Fully active, able to carry on all pre-disease performance without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours.
  Participants
    0 | 14 | 16 | 30
    1 | 90 | 90 | 180
    2 | 11 | 8 | 19
Worst pain score [Count of Participants; unit: Participants] — Pain score range from 0 (no pain) to 10 (pain as bad as you can imagine).
  Participants
    2 | 11 | 12 | 23
    3 | 14 | 19 | 33
    4 | 18 | 15 | 33
    5 | 16 | 18 | 34
    6 | 12 | 14 | 26
    7 | 17 | 10 | 27
    8 | 12 | 11 | 23
    9 | 10 | 5 | 15
    10 | 5 | 10 | 15
Spinal instability neoplastic score (SINS) [Count of Participants; unit: Participants] — SINS is used to assess the stability of the spine in patients with metastatic spinal cord compression. It ranges from 0 to 18; with 0-6 as stable, 7 - 12 as indeterminate and 13-18 instable.
  Participants
    0-6 | 46 | 57 | 103
    > 6 | 69 | 57 | 126
Histology [Count of Participants; unit: Participants]
  Radioresistant | 30 | 30 | 60
  Radiosensitive | 85 | 84 | 169
Mass on imaging [Count of Participants; unit: Participants]
  Absent | 43 | 41 | 84
  Present | 72 | 73 | 145

OUTCOME MEASURES:

1. Primary Outcome: Phase III: Complete Pain Response at 3 Months Post-radiation
Description: A Complete Pain Response is defined as a pain score of zero (0) at the treated site with no concomitant increase in analgesic intake (stable or reducing analgesics in daily oral morphine equivalent) .
Time Frame: 3 months
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Conventional Radiotherapy | Stereotactic Body Radiotherapy
Number analyzed (Participants) | 115 | 114
Participants
  CR | 16 | 40
  PR | 29 | 20
  SD | 34 | 27
  PD | 14 | 7
  In-evalable | 22 | 16
Statistical Analysis 1: Comparison: Standard Conventional Radiotherapy vs Stereotactic Body Radiotherapy; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel — 2-sided, adjusted for stratification factors at randomization; Odds Ratio (OR) = 3.46, 95% CI 2-sided [1.79 to 6.69] — Mantel-Haenszel estimate stratified by stratification factor at randomization

2. Secondary Outcome: Complete Pain Response at 6 Months Post Radiation Based on the International Bone Metastases Consensus Working Party Criteria
Description: as for outcome 1
Time Frame: 6 months post radiation
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Conventional Radiotherapy | Stereotactic Body Radiotherapy
Number analyzed (Participants) | 115 | 114
Participants
  CR | 18 | 37
  PR | 18 | 10
  SD | 32 | 26
  PD | 8 | 5
  In-evaluable | 39 | 36
Statistical Analysis 1: Comparison: Standard Conventional Radiotherapy vs Stereotactic Body Radiotherapy; Test type: Superiority; p = 0.0036, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.56, 95% CI 2-sided [1.35 to 4.85] — Mantel-Haenszel estimate stratified by stratification factors at randomization

3. Secondary Outcome: Radiation Site Progression-free Survival Rate at 6 Months Using MRI Imaging
Description: Radiation site progression was defined as:
  * Gross unequivocal increase in tumor volume or linear dimension > 20%.
  * Any new or progressive tumor within the epidural space.
  * Neurologic deterioration attributable to pre-existing epidural disease with equivocal increased epidural disease dimensions on MRI.
Time Frame: 6 months.
Population: ITT population
Measure: Number (95% Confidence Interval); unit: proportion of participants by arm
Arm/Group | Standard Conventional Radiotherapy | Stereotactic Body Radiotherapy
Number analyzed (Participants) | 115 | 114
proportion of participants by arm | 0.69 [0.60 to 0.77] | 0.75 [0.65 to 0.82]
Statistical Analysis 1: Comparison: Standard Conventional Radiotherapy vs Stereotactic Body Radiotherapy; Test type: Superiority; p = 0.26, Log Rank; 2-sided p-value adjusted for stratification factors at randomization; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.46 to 1.24] — Estimate adjusted for stratification factors at randopmization

4. Secondary Outcome: Overall Survival Rate at 6 Months
Description: Proportion of participants who were alive at 6 months in study.
Time Frame: 6 months post radiation
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: proportion of all participants
Arm/Group | Standard Conventional Radiotherapy | Stereotactic Body Radiotherapy
Number analyzed (Participants) | 115 | 114
proportion of all participants | 0.73 [0.64 to 0.81] | 0.77 [0.68 to 0.84]
Statistical Analysis 1: Comparison: Standard Conventional Radiotherapy vs Stereotactic Body Radiotherapy; Test type: Superiority; p = 0.47, Log Rank — 2-sided p-value adjusted for stratification factors at randomization; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.48 to 1.40]

ADVERSE EVENTS:
Time Frame: 6 months.
Description: Adverse events graded according to CTCAE V4.0
  In the comments, it says that the number of patients in safety analysis does not agree with the patients flow chart. However, they are indeed different. As 115 and 114 were randomized to CRT and SBRT arm respectively, but there were 4 patients on SBRT arm did not receive any treatment, which leads to the difference. (Safety analyses were based on as-treated population)
Arm/Group | Standard Conventional Radiotherapy | Stereotactic Body Radiotherapy
All-Cause Mortality (participants affected / at risk) | 30/115 | 25/114
Serious Adverse Events (participants affected / at risk) | 4/115 | 3/110
Other Adverse Events (participants affected / at risk) | 17/115 | 9/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Conventional Radiotherapy (N=115) | Stereotactic Body Radiotherapy (N=110)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Conventional Radiotherapy (N=115) | Stereotactic Body Radiotherapy (N=110)
Pain (General disorders) | 6 (6) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/65/NCT02512965/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-07): https://cdn.clinicaltrials.gov/large-docs/65/NCT02512965/SAP_001.pdf
  • Informed Consent Form (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/65/NCT02512965/ICF_002.pdf